CLINICAL TRIAL: NCT01677143
Title: Pre-emptive Local Anaesthesia in Gynecological Laparoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SUS2012CMR01; 2012-002356-16 (EudraCT Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-31 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Pain, Postoperative
Keywords: Local anesthetic; Preemptive analgesia; Postoperative pain; Laparoscopy; Gynecological surgery; Day-case surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine (Active Comparator): Injection of 5 ml bupivacaine, 5mg/ml in each port site.
  Interventions: Drug: Bupivacaine 5mg/ml
- Placebo (Placebo Comparator): Injection of 5 ml saline in each port site.
  Interventions: Drug: Bupivacaine 5mg/ml

INTERVENTIONS:
Drug: Bupivacaine 5mg/ml — 5 ml in trocar area
  Other Names: Marcain

SUMMARY:
Pre-emptive local anaesthetics are widely used in laparoscopic surgery, but there is no really consistent evidence that it is useful. Studies in the literature have shown contradicting results. At our hospital we are currently using pre-emptive local anaesthetics in the trocar areas, but as the literature does not give a clear and clinically relevant answer, we need to find out more. This study aims to see if pre-emptive local anaesthetics are useful in the setting of our day-case, laparoscopic surgery.

DETAILED DESCRIPTION:
The study design is prospective, randomized, and double-blinded with parallel assignments. It will compare pre-emptive incisional injection of bupivacaine, 5 mg/ml, with a placebo injection (saline). The clinically relevant comparison should probably be between injection of local anaesthetics and no injection at all. However a study design like that would make blinding impossible and probably not acceptable as a research design for a study which aims to be published.

The aim of the study is to test if pre-emptive injection of long-lasting, local anaesthetics reduces post-operative pain. As local anaesthetics are already implemented in our routine, the hypothesis is that it has a positive effect by reducing postoperative pain. The null hypothesis is that there is no difference between local anaesthetics and placebo.

The recruitment of patients will be from our daily surgery, and consecutive patients who are eligible for day-case, laparoscopic surgery will be asked to participate.

To have a clinically important reduction of post-operative pain a difference of 2 units on a 0-10 numerical rating scale (NRS) is chosen for the sample size calculation. A smaller difference in pain score is not considered clinically relevant in our opinion. With a power of at least 80% this gives 20 patients in total, 10 in each arm. The power calculation was done by statistician S. Johnsen at the University of Surrey. We will include 24 patients altogether to cover for any losses to follow-up. The drop-out rates in clinical trials are usually estimated at 20 %, which would give 25 patients to be included (20/ (1-0.2) = 25). This study has, however, a very short follow-up period, so the drop-out rate is expected to be smaller. Drop-outs will be recorded and accounted for.

24 participants will be randomized in blocks of 6 patients. Block randomization is chosen to avoid pooling by chance.

All procedures will be done by one surgeon. This might be a subject for criticism as one can say that the results in the study are only true for one surgeon in a particular setting. But the need for standardization is very important in studies like this, as pointed out by Wilder-Smith (Wilder-Smith, O. H. 2000).

The time of the randomization is identified as the breakage of the study drug vial. If a potential candidate is found to satisfy any exclusion criteria or withdraws the consent before the vial is opened, the patient is not randomised. The study ID number and the study drug vial will be made available for the next potential candidate.

If a potential candidate is excluded for any reason after the breakage of the vial but before the completion of the injection of the study drug, the study ID number will be coded as Protocol Violation and excluded from the statistical analyses.

The patient, nursing staff and the surgeon will all be blinded to the substance injected.

Infiltration in the primary, umbilical site will be blind, but as close to the fascia as possible. The secondary port infiltrations will be done under visual guidance from the laparoscope, in the fascia and close to the peritoneum. Bupivacaine in a concentration of 5 mg/ml will be used and 5 ml of the solution will be injected at each port site. The patients who get placebo will get 5 ml of physiologic saline injected at each port site.

The primary outcome of the study will be movement-evoked pain (MEP) 5 hours after surgery, as half-life of bupivacaine is 4-6 hours. Movement-evoked pain is the most important outcome measure, because the goal is to get the patient back to normal, daily activities as soon as possible. Trials measuring both movement evoked pain and pain at rest (PAR) suggests that MEP is much more intense than PAR postoperative (Srikandarajah et al, 2011). Pain will be measured on a 10 cm long Numerical Rating Scale (NRS) where 0 cm is no pain and 10 cm is severe pain. NRS is validated as a good tool for pain measurement at different ages and education levels (Gagliese et al, 2005).

Secondary outcome measures will be pain at rest at 2 and 5 hours postoperative, and use of rescue analgesics. Pain at rest must, of course, be recorded before movement evoked pain.

The pain scoring will be done by the patient with help from the nurses at the ward at 2 and 5 hours postoperative, and both will be blinded to which arm the patient is in.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age
* Planned day-case laparoscopic surgery
* Signed Written Informed Consent

Exclusion Criteria:

* ASA score 3-6
* Chronic pain/ Regular use of analgesics
* Inability to understand Norwegian language
* Drug or alcohol abuse
* Inability to understand or sign the Written Informed Consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Postoperative movement-evoked pain | 5 hours postoperative
  The primary outcome of the study will be movement-evoked pain (MEP) 5 hours after surgery, as half-life of bupivacaine is 4-6 hours. Movement-evoked pain is the most important outcome measure, because the goal is to get the patient back to normal, daily activities as soon as possible.

SECONDARY OUTCOMES:
Pain at rest | 2 and 5 hours postoperative
  Secondary outcome measures will be pain at rest at 2 and 5 hours postoperative.
Rescue analgetics | 5 hours postoperative
  Use of rescue analgesics postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Ravndal, MD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway